CLINICAL TRIAL: NCT04200729
Title: Povidone-iodine Irrigation for Prevention of Intra-abdominal Abscess in Pediatric Perforated Appendicitis
Brief Title: Povidone-iodine Irrigation for Prevention of Intra-abdominal Abscess in Pediatric Perforated Appendicitis: a Multi-center Stepped Wedge Cluster Randomized Study
Acronym: PAPPA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, KuoJen Tsao, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HSC-MS-19-0810
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Acute, Perforated Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Therapeutic Irrigation

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomized trial (SW-CRT). After a period of baseline data collection, clusters will be randomized to cross over from control to intervention in a stepwise fashion until all clusters have been exposed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Irrigation with PVI (Experimental)
  Interventions: Drug: Irrigation with PVI
- Usual care (Active Comparator)
  Interventions: Procedure: Usual care

INTERVENTIONS:
Drug: Irrigation with PVI — The intervention will be irrigation with PVI, diluted to a concentration of 1% (containing 0.1% active iodine). After removal of the appendix from the patient's abdomen and attainment of hemostasis,10 mL/kg of 1% PVI solution will be used to irrigate the pelvis and right upper and lower quadrants. The solution will be left to dwell for 1 minute and then suctioned.
  Arms: Irrigation with PVI
Procedure: Usual care — The control will be usual care, which is expected to vary between institutions. The only stipulation for usual care will be that surgeons do not change their usual practice during the baseline period. Some surgeons utilize intra-abdominal irrigation while others use only local irrigation. Intraabdominal irrigation is defined as intraoperative instillation of a large volume (> 200 mL) of irrigation solution into all 4 quadrants of the abdomen. Local irrigation is defined as instillation of a small volume of liquid, typically <50 mL, in the operative field. Intra-abdominal irrigation is utilized with the intention of preventing IAAs while local irrigation is often used to confirm hemostasis or assist with suctioning thick purulent fluid.
  Arms: Usual care

SUMMARY:
The purpose of this study is to determine the effect of intra-abdominal irrigation with povidone-iodine (PVI) versus usual care on the rate of 30-day postoperative intra-abdominal abscesses (IAA) and to determine the effect of PVI irrigation versus usual care on 30-day hospital length of stay(LOS) and 30-day readmissions.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to a participating center
* Appendectomy performed for acute appendicitis
* Intraoperative diagnosis of perforated appendicitis

Exclusion Criteria:

* Simple or gangrenous appendicitis
* Interval or incidental appendectomy
* Initial attempt at non-operative management (defined as >48 hours between the time of diagnosis and surgical intervention)
* History of iodine allergy, thyroid disease or renal dysfunction
* Pregnancy

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1750 (Estimated)
Dates: Start 2027-03-01 (Estimated); Primary Completion 2030-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
number of patients with post operative intra-abdominal abscesses | 30 days post surgery
  An IAA will be defined as: an image-confirmed (ultrasound, CT, or MRI) fluid collection deemed to be an IAA by an attending radiologist or pediatric surgeon, or an abscess confirmed during percutaneous intervention (aspiration of purulent fluid) or reoperation (direct visualization of purulent fluid).

SECONDARY OUTCOMES:
Length of hospital stay(LOS) | 30 days post surgery
  Total 30-day LOS will be defined as the aggregate of all days during which the patient is admitted to the hospital,including any related readmissions, within 30 postoperative days.
Number of patients that are readmitted | 30 days post surgery
  Readmissions will be considered to be related to the index encounter if they are due to abdominal pain, gastrointestinal symptoms, wound related concerns (such as superficial or deep surgical site infection or wound dehiscence), or infection of any kind (such as urinary tract infection, respiratory infection, or symptoms of infection, including fever).

CONTACTS AND LOCATIONS:
Overall Officials: Kuojen Tsao, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No